CLINICAL TRIAL: NCT06732804
Title: A Randomised, Parallel Group Treatment, Double-blind, 3-arm Study to Investigate the Comparative PK, Safety, Immunogenicity, and Tolerability Between AVT80 and Entyvio® in Healthy Male and Female Participants Aged 18 to 55 Years Inclusive
Brief Title: Study to Investigate Comparative Pharmacokinetics, Safety, Immunogenicity and Tolerability Between AVT80 and Entyvio
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVT80-GL-P01
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Male and Female Subjects
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AVT80 (Experimental): Single subcutaneous administration of AVT80
  Interventions: Biological: AVT80
- Geographical region 1 Entyvio (Active Comparator): Single subcutaneous administration of Geographical region 1 Entyvio
  Interventions: Biological: Geographical region 1 Entyvio
- Geographical region 2 Entyvio (Active Comparator): Single subcutaneous administration of Geographical region 2 Entyvio
  Interventions: Biological: Geographical region 2 Entyvio

INTERVENTIONS:
Biological: AVT80 — Single subcutaneous injection of AVT80 (108mg)
  Arms: AVT80
Biological: Geographical region 1 Entyvio — Single subcutaneous injection of Geographical region 1 Entyvio (108mg)
  Arms: Geographical region 1 Entyvio
Biological: Geographical region 2 Entyvio — Single subcutaneous injection of Geographical region 2 Entyvio (108mg)
  Arms: Geographical region 2 Entyvio

SUMMARY:
The study has been designed as a randomised, parallel-group, double-blind, 3 arm study to investigate the comparative pharmacokinetics, safety, immunogenicity and tolerability between AVT80 and Entyvio in healthy volunteers.

DETAILED DESCRIPTION:
The study will consist of a screening period, a treatment and assessment period and an End of Study visit. Eligibility for the study will be determined during a screening period. Subjects who meet the eligibility criteria will be randomised to receive a single dose of either AVT80, geographical region 1 Entyvio or geographical region 2 Entyvio.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participant capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in the protocol.
* Have a body weight of 50.0 to 90.0 kg (inclusive) and body mass index (BMI) of 17.0 to 32.0 kg/m2 (inclusive).
* Participant must be 18 to 55 years old inclusive, at the time of signing the ICF.

Exclusion Criteria:

* Participant has a history of relevant drug and/or food allergies.
* Participant has a history of hypersensitivity to Entyvio, AVT80, or their constituents.
* Participant has any past or concurrent medical conditions that could potentially increase the participant's risks or that would interfere with the study evaluation, procedures, or study completion. Examples of these include medical history with evidence of clinically relevant pathology (e.g., demyelinating disorders).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 385 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate PK similarity of AVT80 with geographical region 1 Entyvio and geographical region 2 Entyvio and between geographical region 1 Entyvio and geographical region 2 Entyvio | Day Zero to Day 126
  PK endpoint of Cmax.
To demonstrate PK similarity of AVT80 with geographical region 1 Entyvio and geographical region 2 Entyvio and between geographical region 1 Entyvio and geographical region 2 Entyvio | Day Zero to Day 126
  PK endpoint of AUC0-inf.

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Schurink, Study Director — Alvotech Swiss AG
Locations (3):
- Veritus Research Pty Ltd, Bayswater, Australia
- New Zealand (2):
  - Investigational Site 0002, Auckland
  - NZCR, Christchurch

IPD SHARING:
Plan to Share IPD: No